CLINICAL TRIAL: NCT07113119
Title: Effects of a Long-term Exercise Training Program on the Functional Capacity and Health-related Quality of Life in Inpatients With Psychotic Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor of Sports Medicine, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EH-44/2021
Record Dates: First submitted 2025-07-30; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Psychotic Disorder
Keywords: Exercise; Functional ability; Quality of life; Pilates
MeSH Terms: conditions — Psychotic Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A: EXERCISE GROUP (Experimental): Exercise group: 1-year mixed-type exercise training program
  Interventions: Other: Exercise intervention
- GROUP B: CONTROL GROUP (No Intervention): Control Group: 1-year normal physical activity, without participating in organized sports programs

INTERVENTIONS:
Other: Exercise intervention — Patients that will be randomly assigned in the group A will be invited to attent 1-year exercise sessions, with frequency 3 sessions per week. The program included 30 minutes of Pilates exercises, strengthening, balance and flexibility exercises, which are performed with rubber bands, mobility sticks and balls.
  Arms: GROUP A: EXERCISE GROUP

SUMMARY:
Mental health represents a fundamental dimension of overall well-being, exerting a significant influence on mortality rates, health-related quality of life (HRQoL), levels of disability, and the strain on healthcare systems. As the interest in mental wellness continues to grow, exercise training (ET) has become increasingly recognized as a validated and effective intervention for individuals experiencing mental health challenges. An expanding body of research underscores the adverse effects of physical inactivity, reinforcing the role of exercise as a viable therapeutic strategy.

Well-structured ET interventions have consistently demonstrated benefits across multiple domains, including improvements in physical health, reductions in cardiovascular risk, and enhancements in psychological constructs such as depression, self-esteem, resilience, and self-efficacy. However, the majority of prior studies have been limited to relatively short durations-typically ranging from 4 to 24 weeks, with an average of about 12 weeks. A significant gap in the literature persists regarding the long-term implementation and effectiveness of ET programs, particularly in populations with severe mental illness. Additionally, the small sample sizes commonly seen in previous studies restrict the statistical robustness and generalizability of their outcomes.

The aim of the randomized control trial is to examine whether an 1-year mixed type exercise training program within the hospital setting will improve functional capacity and health-related quality of life. Forty- eight participants will be randomly allocated into two groups: Group A (Exercise group) will receive 3 exercise sessions per week for 1-year and Group B (Control Group) will continue their usual care, without participating in organized exercise programs. Prior to the group random allocation, part of the assessment at the baseline and 1 year follow-up will include lower extremity strength test, muscle power using a dynamometer, aerobic capacity test, balance test, body positioning and health- related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* being an adult
* inpatient with a diagnosis of psychotic syndrome
* on stable medication
* controlled as far as psychosis is concerned
* consenting to participate

Exclusion Criteria:

* adolescents
* with other diagnoses
* not on stable medication
* in an unstable condition
* unwilling to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-08-04 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Isometric Lower Extremity Strength Assessment in Semi-Squat Using Baseline Leg Dynamometer | Baseline
  The isometric strength of the lower extremities is evaluated in a semi-squat position using a Baseline Leg Dynamometer, with musclular strength quantified in kilograms (kg).
Isometric Lower Extremity Strength Assessment in Semi-Squat Using Baseline Leg Dynamometer | Follow-up assessment, 12 months post- baseline
  The isometric strength of the lower extremities is evaluated in a semi-squat position using a Baseline Leg Dynamometer, with muscular strength quantified in kilograms (kg).
Handgrip Strength | Baseline
  Evaluation of the isometric handgrip strength using a hand dynamometer
Handgrip Strength | Follow-up assessment, 12 months post- baseline
  Evaluation of the isometric handgrip strength using a hand dynamometer
Sit-and-Reach Test | Baseline
  Evaluation of flexibility using sit- and- reach test
Sit-and-Reach Test | Follow-up assessment, 12 months post- baseline
  Evaluation of flexibility using sit- and- reach test
30 -second Sit-to-stand test (STS) | Baseline
  Evaluation of functional capacity and mobility using 30-second STS
30 -second Sit-to-stand test (STS) | Follow-up assessment, 12 months post- baseline
  Evaluation of functional capacity and mobility using 30-second STS
Six- Minute Walking Test | Baseline
  Estimation of aerobic capacity through six minute walking test
Six- Minute Walking Test | Follow-up assessment, 12 months post- baseline
  Estimation of aerobic capacity through six minute walking test
Berg Balance Scale Test | Baseline
  Evaluation of balance using Berg Balance Scale Test
Berg Balance Scale Test | Follow-up assessment, 12 months post- baseline
  Evaluation of balance using Berg Balance Scale Test
Short form Quality of Life (SF-36) | Baseline
  Assessment of Quality of Life using SF-36
Short form Quality of Life (SF-36) | Follow-up assessment, 12 months post- baseline
  Assessment of Quality of Life using SF-36

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Medicine Laboratory, Aristotle University of Thessaloniki, Thessaloniki, Thermi, Greece